CLINICAL TRIAL: NCT03954236
Title: A Pilot, Prospective, Randomized, Double-Blinded, Vehicle- and Comparator-Controlled Trial on Safety and Efficacy of a Topical Inhibitor of Janus Kinase 1/2 (Ruxolitinib INCB018424 Phosphate 1.5% Cream) for Non-Sclerotic Chronic Cutaneous Graft-Versus-Host Disease
Brief Title: Study of the Safety and Efficacy of Ruxolitinib Cream for Non-Sclerotic Chronic Cutaneous Graft-Versus-Host Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hackensack Meridian Health (Other); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-412
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Non-sclerotic Cutaneous Chronic Graft-versus-host Disease
Keywords: Ruxolitinib Cream; 18-412
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with graft-versus-host disease (GVHD) (Experimental): Participants will have non-sclerotic chronic cutaneous graft-versus-host disease (GVHD) or you have a condition called superficially sclerotic chronic cutaneous graft-versus-host disease (GVHD) after having received an allogeneic hematopoietic stem cell transplant.
  Interventions: Drug: topical ruxolitinib 1.5% cream; Other: Topical vehicle/moisturizer cream

INTERVENTIONS:
Drug: topical ruxolitinib 1.5% cream — Patients will be prescribed twice daily use of topical ruxolitinib 1.5% cream (randomized half of face/body) to a maximum of 20% BSA on each side for 28 ± 3 days. Topical ruxolitinib will be provided as topical cream. At the end of the 28 ± 3 days study visit, patients will remain blinded to treatment arms. After trial completion (day 28 ± 3 days), all patients will be offered repeated treatment cycle with topical ruxolitinib or standard of care therapy.
Other: Topical vehicle/moisturizer cream — Patients will be prescribed twice daily use of vehicle/moisturizer (for contralateral side of face/body) to a maximum of 20% BSA on each side for 28 ± 3 days.At the end of the 28 ± 3 days study visit, patients will remain blinded to treatment arms. After trial completion (day 28 ± 3 days), all patients will be offered repeated treatment cycle with topical ruxolitinib or standard of care therapy.

SUMMARY:
The purpose of this study is to compare the safety and effects of ruxolitinib 1.5% cream with those of standard moisturizers in people with non-sclerotic chronic cutaneous GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥ 12 years)
* History of allogeneic hematopoietic stem cell transplantation
* BSA of at least 2% of clinically or histologically confirmed non-sclerotic cutaneous chronic graft-versus-host disease (diagnosed and BSA calculated in accordance with the National Institutes of Health Chronic Graft-versus-Host Disease Consensus for Clinical Trials: I. The 2014 Diagnosis and Staging Working Group Report)
* Patients age ≥ 18 years must provide written informed consent; or patients age ≥12 years and <18 years must provide assent and have at least one guardian provide written informed consent to participate in the study.
* Able to self-administer topical interventions or provide for another person to apply the topical interventions (while wearing nitrile gloves)
* If on systemic therapy for GVHD, systemic therapy must be stable for past 4 weeks; however, any planned systemic corticosteroid taper during the study will be permitted.Changes in systemic therapy during the study period will be allowed for the management of non-skin GVHD.
* Any concurrent topical therapies including topical corticosteroids, topical calcienurin inhibitors, moisturizers, phototherapy (narrowband UVB or UVA1); or excimer laser therapy must be discontinued on Study Day 0.

Exclusion Criteria:

* Known history of allergy to any ingredient of the study medication
* Patients with deep sclerotic cutaneous graft-versus-host disease including deep sclerotic subtypes of chronic cutaneous GVHD
* Use of concurrent topical therapy including topical corticosteroids, topical calcienurin inhibitors, moisturizers, phototherapy (narrowband UVB or UVA1); or excimer laser therapy after Study Day 0 up to and including Study Day 28.
* Changes in systemic therapy during study period for the purpose of treating skin GVHD.
* Special populations:

  * vulnerable populations e.g. decisionally impaired (cognitive, psychiatric), terminally ill, prisoners
  * patients who, in the opinion of the investigator have a condition that precludes their ability to provide an informed consent
* Concurrent participation in another topical trial of a drug(s) or medical device, or the subject is in an exclusion period after a previous trial of drug(s) or medical device
* Pregnancy or lactation
* Patients with inadequate liver function (ALT above 4 × upper limit of normal [ULN] for the patient's age or direct bilirubin 4 × ULN for the patient's age and the laboratory abnormalities are considered to be due to underlying liver dysfunction) unless attributed to GVHD (if direct bilirubin is not in the medical record, it is acceptable to use total bilirubin x4 ULN).
* Active uncontrolled infection requiring systemic therapy. Subjects with a controlled infection receiving definitive therapy for 48 hours prior to enrollment are eligible.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2027-02-06 (Estimated); Study Completion 2027-02-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Participants With Graft-versus-host Disease (GVHD): Topical ruxolitinib BID to left side of face/body, And topical moisturizer BID to right side of face/body
- Group 2: Participants With Graft-versus-host Disease (GVHD): Topical ruxolitinib BID to right side of face/body And topical moisturizer BID to left side of face/body
Period: Overall Study
Arm/Group | Group 1: Participants With Graft-versus-host Disease (GVHD) | Group 2: Participants With Graft-versus-host Disease (GVHD)
Started | 12 | 12
Completed | 10 | 10
Not Completed | 2 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Ruxolitinib treatment plan assigned
Groups:
- Experimental: Participants With Graft-versus-host Disease (GVHD): All Study Participants: topical ruxolitinib BID to one side of face/body
Arm/Group | Experimental: Participants With Graft-versus-host Disease (GVHD)
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 52 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Body Surface Area (BSA) From Day 1 and Day 28
Description: The difference in BSA of non-sclerotic cutaneous cGVHD between ruxolitinib treated side and vehicle treated sides of the face/body at study completion
Time Frame: 28 days (+/-3 days)
Population: 12 participants were assessed for each grouping of interventions
Measure: Mean (Standard Error); unit: % of body surface area
Arm/Group | Experimental: Participants With Graft-versus-host Disease (GVHD)
Number analyzed (Participants) | 24
% of body surface area
  BSA on Day 1 for Topical Ruxolitinib BID to Left Side of Face/Body: number analyzed (Participants) | 12
  BSA on Day 1 for Topical Ruxolitinib BID to Left Side of Face/Body | 14.4 (0.003)
  BSA on Day 28 for Topical Ruxolitinib BID to Left Side of Face/Body: number analyzed (Participants) | 12
  BSA on Day 28 for Topical Ruxolitinib BID to Left Side of Face/Body | 6.2 (0.003)
  BSA on Day 1 for Topical Ruxolitinib BID to Right Side of Face/Body: number analyzed (Participants) | 12
  BSA on Day 1 for Topical Ruxolitinib BID to Right Side of Face/Body | 14.5 (0.003)
  BSA on Day 28 for Topical Ruxolitinib BID to Right Side of Face/Body: number analyzed (Participants) | 12
  BSA on Day 28 for Topical Ruxolitinib BID to Right Side of Face/Body | 10.4 (0.003)

2. Secondary Outcome: Improvement in Physician's Global Assessment of Clinical Condition (PGA) at From Day 1 and Day 28
Description: The difference in the Physician's Global Assessment/PGA of non-sclerotic and superficially sclerotic cutaneous cGVHD between ruxolitinib treated side and vehicle treated sides of the face/body at study completion (day 28 visit). Grade of Rash as follows: Grade 0, Clinical Complete Response, Completely clear; NED (100% improvement); Grade 1-3, Partial Response, from very significant clearance to moderate improvement (>90% to >/= 50% improvement); Grade 4 and 5, Stable Disease, No change to some improvement (,50% to >/=25%); Grade 6, Progressive Disease, Disease is worse than at baseline evaluation by >/= 25%.
Time Frame: 28 days (+/-3 days)
Population: 12 participants were assessed for each grouping of interventions
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Participants With Graft-versus-host Disease (GVHD)
Number analyzed (Participants) | 24
units on a scale
  Topical Ruxolitinib BID to Left Side of Face/Body PGA on Day 1: number analyzed (Participants) | 12
  Topical Ruxolitinib BID to Left Side of Face/Body PGA on Day 1 | 5 (0.0004)
  Topical Ruxolitinib BID to Left Side of Face/Body PGA on Day 28: number analyzed (Participants) | 12
  Topical Ruxolitinib BID to Left Side of Face/Body PGA on Day 28 | 1.9 (0.0004)
  Topical Ruxolitinib BID to Right Side of Face/Body PGA on Day 1: number analyzed (Participants) | 12
  Topical Ruxolitinib BID to Right Side of Face/Body PGA on Day 1 | 5 (0.0004)
  Topical Ruxolitinib BID to Right Side of Face/Body PGA on Day 28: number analyzed (Participants) | 12
  Topical Ruxolitinib BID to Right Side of Face/Body PGA on Day 28 | 3.7 (0.0004)

ADVERSE EVENTS:
Time Frame: 28 days (+/-3 days)
Groups:
- Experimental Left: Participants With Graft-versus-host Disease (GVHD): topical ruxolitinib BID to left side of face/body
- Experimental Right: Participants With Graft-versus-host Disease (GVHD): topical ruxolitinib BID to right side of face/body
Arm/Group | Experimental: Participants With Graft-versus-host Disease (GVHD) | Experimental Left: Participants With Graft-versus-host Disease (GVHD) | Experimental Right: Participants With Graft-versus-host Disease (GVHD)
All-Cause Mortality (participants affected / at risk) | 8/24 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/24 | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Participants With Graft-versus-host Disease (GVHD) (N=24) | Experimental Left: Participants With Graft-versus-host Disease (GVHD) (N=12) | Experimental Right: Participants With Graft-versus-host Disease (GVHD) (N=12)
Sinusitis (Infections and infestations) | 1 | 0 | 0
Neoplasm Benign, Malignant and Unspecified (incl cysts and polyps) - Other, specify - CNS Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Participants With Graft-versus-host Disease (GVHD) (N=24) | Experimental Left: Participants With Graft-versus-host Disease (GVHD) (N=12) | Experimental Right: Participants With Graft-versus-host Disease (GVHD) (N=12)
Sinusitis (Infections and infestations) | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Cracked/thick cuticles (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Nummular eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Orofacial dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Eyelash hypotrichosis (Eye disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT03954236/Prot_SAP_000.pdf